CLINICAL TRIAL: NCT03706482
Title: An Exploratory, Open Label, Multiple Dose, Multicentre Phase I/II Trial Evaluating Safety and Efficacy of Postnatal or Prenatal and Postnatal Intravenous Administration of Allogeneic Expanded Fetal Mesenchymal Stem Cells for the Treatment of Severe Osteogenesis Imperfecta Compared With a Combination of Historical and Untreated Prospective Controls
Brief Title: Boost Brittle Bones Before Birth
Acronym: BOOSTB4
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University College, London (Other); Universitätsklinikum Köln (Other); UMC Utrecht (Other); Leiden University Medical Center (Other); Lund University (Other)
Responsible Party: Principal Investigator, Cecilia Götherström, Sponsor's representative, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIBB01; 2015-003699-60 (EudraCT Number)
Record Dates: First submitted 2018-10-05; First posted 2018-10-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Postnatal (Experimental): 15 participants.
  Administration of four postnatal doses of BOOST cells with the first dose as soon as possible after birth and the three additional doses at +4, +8 and +12 months after the first dose. Each dose is 3x10^6 MSC/kg body weight.
  Interventions: Biological: BOOST cells
- Prenatal (Experimental): 3 participants.
  Administration of one prenatal dose of BOOST cells followed by three postnatal doses at +4, +8 and +12 months after the first dose. Each dose is 3x10^6 MSC/kg body weight.
  Interventions: Biological: BOOST cells
- Prospective control (untreated) (No Intervention): 1-30 participants.
  Subjects eligible for the trial but not willing/able to participate in any of the experimental arms.
- Historic control (No Intervention): 18-90 participants (1-5 per included and treated subject).
  Matched historical controls. Subjects will be identified in historical registries and data will be retrieved from national OI registers and the OI Variant Database (Dalgleish 2018).

INTERVENTIONS:
Biological: BOOST cells — Four doses of expanded human 1st trimester fetal liver-derived mesenchymal stem cells.
  Arms: Postnatal; Prenatal

SUMMARY:
An exploratory, open label, multiple dose, multicentre phase I/II trial evaluating safety and efficacy of postnatal or prenatal and postnatal administration of allogeneic expanded fetal mesenchymal stem cells for the treatment of severe Osteogenesis Imperfecta compared with a combination of historical and untreated prospective controls.

ELIGIBILITY:
Inclusion Criteria Postnatal Group:

1. Parent's/legal guardian's signed informed-consent form
2. Clinical diagnosis of OI type III or severe type IV AND
3. Molecular diagnosis of OI (Glycine substitution in the collagen triple-helix encoding region of either the COL1A1 or COL1A2 gene)
4. Age less than 18 months (calculated from gestational week 40+0, i.e. the corrected age)
5. Parent/legal guardian over 18 years of age

Inclusion Criteria Prenatal Group:

1. Woman has signed the informed-consent form
2. Only women where termination of the pregnancy is no longer possible or where the women are committed to continue the pregnancy may be included in the trial
3. Suspicion of OI type III or severe type IV in the fetus on ultrasound findings AND
4. Molecular diagnosis of OI in the fetus (Glycine substitution in the collagen triple-helix encoding region of either the COL1A1 or COL1A2 gene)
5. Gestation age between 16+0 and 35+6 weeks+days
6. Pregnant woman over 18 years of age

Inclusion Criteria Historical Control Group:

1. Parent's/legal guardian's signed informed-consent form
2. Clinical and molecular diagnosis of OI (Glycine substitution in the collagen triple-helix encoding region of either the COL1A1 or COL1A2 gene)
3. Data on fractures and growth is available
4. Parent/legal guardian over 18 years of age

Inclusion Criteria Prospective Untreated Control Group:

* Postnatal inclusion: The inclusion criteria for the postnatal group apply.
* Prenatal inclusion: The inclusion criteria for the prenatal group apply, except inclusion criteria 2.

Exclusion Criteria Postnatal Group:

1. Existence of other known disorder that might interfere with the treatment, such as, but not limited to organ dysfunction (for example liver or renal failure or bronchopulmonary dysplasia), congenital heart defect, hypoxic encephalopathy l-lll, severe neurological problems, immune deficiencies, muscle diseases, severe malformations or syndromes diagnosed by clinical examination.
2. Any contraindication for invasive procedures such as a moderate/severe bleeding tendency
3. Known risk factors for clotting, such as, but not limited to previous blood clot, family history of clots, clotting disorder (inherited or acquired), heart failure, inflammatory disorders (for example lupus, rheumatoid arthritis, inflammatory bowel disease)
4. Positive Donor Specific Antibody-test
5. Known allergy/hypersensitivity to Fungizone and/or Gensumycin
6. Abnormal karyotype or other confirmed genetic syndromes
7. Oncologic disease (previous or current malignancy)
8. Inability to comply with the trial protocol and follow-up schedule
9. Inability to understand the information and to provide informed consent

Exclusion Criteria Prenatal Group:

1. Multiple pregnancy
2. Co-existence of other disorder that might interfere with the treatment, as judged by the Investigator or the patient's obstetrician
3. Abnormal fetal karyotype or other confirmed genetic syndrome
4. Any contraindication for invasive procedures such as a bleeding tendency or contagious infections, such as, but not limited to HIV, Syphilis, Hepatitis B, Hepatitis C or other known infectious diseases that can harm the fetus
5. Known risk factors for clotting, such as, but not limited to previous blood clot, family history of clots, clotting disorder (inherited or acquired), heart failure, inflammatory disorders (for example lupus, rheumatoid arthritis, inflammatory bowel disease)
6. Positive Donor Specific Antibody-test
7. Known allergy/hypersensitivity to Fungizone and/or Gensumycin
8. Oncologic disease in woman or fetus (previous or current malignancy)
9. Unwilling to or cannot undergo delivery by elective Caesarean section
10. Inability to comply with the trial protocol and follow-up schedule
11. Inability to understand the information and to provide informed consent

Exclusion Criteria Historical Control Group:

1. Existence of other disorder that might interfere with the trial. No lung hypoplasia (type II OI).
2. Abnormal karyotype

Exclusion Criteria Prospective Untreated Control Group:

* Postnatal inclusion: The exclusion criteria, except exclusion criterium 2, 3, 4 and 5 (Contraindication for invasive procedure, Known risk factor for clotting, Positive Donor Specific Antibody-test and Known allergy/hypersensitivity to Fungizone and/or Gensumycin) for the postnatal group apply.
* Prenatal inclusion: The exclusion criteria, except exclusion criterium 1, 4, 5, 6 and 7 (Multiple pregnancy, Contraindication for invasive procedure, Known risk factor for clotting, Positive Donor Specific Antibody-test and Known allergy/hypersensitivity to Fungizone and/or Gensumycin) for the prenatal group apply.

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability measured as seriousness, severity and frequency of treatment related adverse events. | From baseline to the long-time follow-up (10 years after the first dose).
  The primary endpoint is safety and tolerability measured as seriousness, severity and frequency of treatment related adverse events (AEs), with specific focus on the following:
  1. Vital signs in conjunction with the MSC administration
  2. Transfusion reactions (administration toxicity, allergy, embolism)
  3. Immune reaction with or without symptoms of inflammation, potentially resulting in rejection of the cells or development of donor-specific antibodies:
     * Allergy or Hypersensitivity responses to antibiotics or antimycotics
     * Development of Fetal Bovine Serum-specific antibodies
     * Hypersensitivity responses to Human Serum Albumin
     * Hypersensitivity to impurities in the IMP
  4. Prenatal complications (miscarriage/intrauterine fetal death, premature birth, infection in utero or persistent [>1 min] fetal bradycardia) in the prenatal group
  5. Adverse effects of feto-maternal transmission of donor cells in the prenatal group
  6. Tumourigenicity
  7. Mortality/morbidity

SECONDARY OUTCOMES:
Number of fractures. | From baseline to the primary follow-up (6 and 12 months after the last dose) and therafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Number of fractures.
Time (days) to first fracture after each stem cell administration. | From each dose of stem cells to the time point of the first fracture. Assessed up to 10 years after the first stem cell dose.
  Time (days) to first fracture after each stem cell administration.
Numbers of fractures at birth. | Evaluated at birth.
  Numbers of fractures at birth.
Change in bone-marrow density (g/cm2). | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Change in bone-marrow density (g/cm2).
Growth (cm). | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Growth (cm) as assessed by clinician.
Growth (kg). | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Growth (kg) as assessed by clinician.
Change in clinical status of OI. | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Change in clinical status of OI based on parameters defined under efficacy assessments described in protocol, as assessed by OI clinician.
Assessment of biochemical bone turnover by analysis of the markers P-Calcium, P-Phosphate, P-Albumin, S-ALP, fP-PTH, S-25-OH Vitamin D, Bone specific S-ALP, S-CTx, S-Osteocalcin and U-DPD/Krea and U-NTx/Krea in blood and urine samples. | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Assessment of biochemical bone turnover.

OTHER OUTCOMES:
Impact on the subjects Quality of Life: Infant Toddler Quality of Life Questionnaire™ (ITQOL) | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Quality of life assessed using the Infant Toddler Quality of Life Questionnaire™ (ITQOL).
Incidence of donor cells engrafted into patient tissue samples assessed by histology. | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Donor cell engraftment.
Analysis of an array of cytokines and micro vesicles to evaluate paracrine effects. | From baseline to the primary follow-up (6 and 12 months after the last dose) and thereafter assessed annually to the end of the long-time follow-up (10 years after the first dose).
  Paracrine effects will be analysed from plasma isolated from peripheral blood.
Assess the potential of non-invasive methods of prenatal diagnosis for OI by genetic analysis of parent DNA. | From baseline to birth for prenatal group.
  Non-invasive prenatal diagnosis will be studied during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Åström, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this trial, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent ethics review committee can submit proposals up to 36 months following article publication. After 36 months the data will be available in our Institute's data warehouse but without investigator support other than deposited metadata. Since the IPD is coded and a code key exists, study participants can be identified indirectly via the code key and the IPD is classified as personal data according to the GDPR General Data Protection Regulation (Regulation (EU) 2016/679). Data requestors will need to adhere to GDPR and sign a data transfer agreement. Data requestors from non-EU/EES countries will also need to sign the EU commissions Standard Contractual Clauses for data transfer between EU and non-EU countries. Proposals should be directed to boostb4@clintec.ki.se.
URL: http://www.boostb4.eu

REFERENCES:
- [Derived] Sagar RL, Astrom E, Chitty LS, Crowe B, David AL, DeVile C, Forsmark A, Franzen V, Hermeren G, Hill M, Johansson M, Lindemans C, Lindgren P, Nijhuis W, Oepkes D, Rehberg M, Sahlin NE, Sakkers R, Semler O, Sundin M, Walther-Jallow L, Verweij EJTJ, Westgren M, Gotherstrom C. An exploratory open-label multicentre phase I/II trial evaluating the safety and efficacy of postnatal or prenatal and postnatal administration of allogeneic expanded fetal mesenchymal stem cells for the treatment of severe osteogenesis imperfecta in infants and fetuses: the BOOSTB4 trial protocol. BMJ Open. 2024 Jun 4;14(6):e079767. doi: 10.1136/bmjopen-2023-079767. PMID 38834319